CLINICAL TRIAL: NCT01435525
Title: Nexium Capsules Specific Clinical Experience Investigation Concerning Helicobacter Pylori Eradication
Brief Title: Nexium Capsules Helicobacter Pylori Specific Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961HC00011
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Gastric Ulcer; Duodenal Ulcer; Gastric Mucosa-associated Lymphoid Tissue (MALT); Lymphoma Idiopathic Thrombocytopenic Purpura; Early Gastric Cancer
Keywords: triple therapy; Helicobacter pylori; eradication; Nexium
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nexium

SUMMARY:
The purpose of this study is to confirm the safety profile / factors which impact safety and efficacy in patients given triple therapy for Helicobacter pylori eradication with Nexium + amoxicillin (AMPC) + clarithromycin (CAM), or Nexium + AMPC + metronidazole (MNZ) in usual post-marketing use.

DETAILED DESCRIPTION:
Nexium capsules Specific Clinical Experience Investigation concerning Helicobacter pylori eradication

ELIGIBILITY:
Inclusion criteria:

* Triple therapy for H.pylori eradication to stomach started after endoscopic treatment for gastric ulcer
* Triple therapy for H.pylori eradication to stomach started after endoscopic treatment for duodenal ulcer
* Triple therapy for H.pylori eradication to stomach started after endoscopic treatment for gastric MALT lymphoma
* Triple therapy for H.pylori eradication to stomach started after endoscopic treatment for idiopathic thrombocytopenic purpura
* Triple therapy for H.pylori eradication to stomach started after endoscopic treatment for early gastric cancer

Exclusion Criteria:

- H.pylori negative at the time when the triple therapy is started

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients to whom triple therapy for H.pylori eradication to stomach is started after endoscopic treatment for gastric ulcer, duodenal ulcer, gastric MALT lymphoma, idiopathic thrombocytopenic purpura, or early gastric cancer as the approved indication of Nexium. Patients with H.pylori negative at the time when the triple therapy is started are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Drug Reactions | Period from the start of triple therapy to assessment of eradication, an expected average of 3 months

SECONDARY OUTCOMES:
Rate of H.Pylori eradication | Period from the start of triple therapy to assessment of eradication, an expected average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (36):
- Japan (36):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamanashi